CLINICAL TRIAL: NCT03868202
Title: Follicle Stimulating Hormone (FSH) Glycosylation in Women: Effect of Estradiol
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: Wichita State University (Other)
Responsible Party: Principal Investigator, Reem Sabouni, Principal Investigator, Fellow of Reproductive Endocrinology and Infertility, Eastern Virginia Medical School
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 19-03-FB-0058-EVMS
Record Dates: First submitted 2019-03-04; First posted 2019-03-11 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Follicle Stimulating Hormone Glycosylation; Urinary FSH21/FSH24 Ratio; Estradiol Effect
MeSH Terms: interventions — Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Premenopausal women (No Intervention): Participants will bring into clinic their first voided urine of the day on cycle days 9, 12 and 15 in a urinary collection kit that will be given. A urine dip stick will be performed on the samples. Each time they bring in a sample, they will have a serum blood draw for estradiol and FSH.
- Postmenopausal women (Active Comparator): Participants will bring into clinic their first voided urine of the day on assigned days 1, 4 and 7 in a urinary collection kit that will be given. A urine dip stick will be performed on the samples. Each time they bring in a sample, they will have a serum blood draw for estradiol and FSH. The participants will then be started on EstroGel© for 14 days from day 7-21. During that time that they are on EstroGel©, the participants will bring into clinic their first voided urine of the day on assigned days 15, 18, and 21 in a urinary collection kit that will be given. A urine dip stick will be performed on the samples. Each time they bring in a sample, they will have a serum blood draw for estradiol and FSH. After the last urinary collection and blood draw, they will discontinue the EstroGel and be started on micronized progesterone if they have a uterus for 12 days.
  Interventions: Drug: Estradiol Transdermal Product

INTERVENTIONS:
Drug: Estradiol Transdermal Product — Hormone replacement therapy will be given to postmenopausal women for up to 1 month.
  Other Names: Micronized progesterone
  Arms: Postmenopausal women

SUMMARY:
This clinical trial is an investigational research study to determine the ratio of glycosylated FSH21/FSH24 in premenopausal women and postmenopausal women as well as determining if estradiol can increase this ratio in postmenopausal women.

DETAILED DESCRIPTION:
Follicle Stimulating Hormone (FSH), is secreted by the pituitary gland at the base of the brain, and is the primary stimulus for growth of the ovarian follicle that contains the egg. Glycosylation, or adding glucose, to FSH is critical for its bioactivity on stimulating the ovarian follicle. The FSH with less glycosylation (FSH21) has a higher affinity for the FSH receptor and activates more pathways than does fully-glycosylated FSH (FSH24). Previous studies showed pituitaries from young women contain a high ratio of FSH21/FSH24 while pituitaries from older and postmenopausal women have a lower ratio of FSH21/FSH24. The investigators hypothesize that the higher FSH21/FSH24 ratio found in young women is responsible for normal follicle growth.

This study is intended to provide the first determination of systemic changes in the ratio of FSH21/FSH24 and determine if estradiol increases the FSH21/FSH24 ratio in the first morning urine of women. To take part in this study, the participant must be willing to collect the first morning urine on particular mornings of the menstrual cycle and be available for blood draws on those mornings. Additionally for postmenopausal participants, the participant must be willing to use topical estrogen, EstroGel©, for 14 days and be willing to collect the first morning urine on particular mornings and again be available for blood draws on those mornings. For the postmenopausal participants with an intact uterus, the participants must be willing to take an oral progestin, micronized progesterone, for 12 days following the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

Premenopausal (Age 20-30):

1. Age between 20 - 30 years old
2. Not on oral, transdermal or vaginal hormonal contraception with last use greater than 2 months (non-hormonal IUD okay)
3. At least 6 weeks after removal of subdermal contraceptive implant
4. At least 9 months from the last hormonal contraceptive injection
5. Regular menses with a 26-32 day interval
6. Willingness to abstain from heterosexual intercourse or use barrier contraception during the study
7. No serious medical illness
8. Not on medication(s) effecting ovarian function
9. Screening ultrasound on cycle day 12-14 with at least 1 follicle measuring >12mm.
10. Normal pap smear within the last 3 years, if indicated (report needed)

Postmenopausal (Age 45-60):

1. Age between 45-60 years old
2. Last spontaneous menstrual period >1 year
3. Vaginal pH > 5.0
4. No contraindications to hormonal replacement therapy
5. No major medical condition/current medication(s) that would impact use of hormone replacement therapy
6. Never have been on hormone replacement therapy or last use greater than 6 months
7. Mammogram within the last 1 year that is normal (report needed)
8. Pap smear within the last 3-5 years that is normal (report needed)
9. Willing to use hormone replacement therapy

Exclusion Criteria:

Premenopausal (Age 20-30):

1. Uncorrected endocrinopathy affecting ovarian function (i.e.: Prolactinoma, thyroid disease)
2. Medications affecting the hypothalamic-pituitary-ovarian axis.
3. Screening ultrasound with no follicles measuring ≥11 mm
4. History of pelvic surgery
5. Current abnormal pap smear requiring intervention

Postmenopausal (Age 45-60):

1. Last menstrual period <1 year
2. Contraindication to hormone replacement therapy
3. Use of exogenous hormone replacement therapy in the last 6 months
4. Significant medical disease or current medication use that can impact estrogen metabolism
5. Unwilling or unable to use transdermal estrogen and oral progestin.
6. Allergy to transdermal estrogen and oral progestin.
7. Unexplained vaginal bleeding within the last 6 months.

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-07-03 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
The ratio of urinary FSH21/FSH24 and total FSH levels in urine of young women versus postmenopausal women. | up to 4 weeks for each participant
The levels of serum estradiol and FSH in young women versus postmenopausal women. | up to 4 weeks for each participant

CONTACTS AND LOCATIONS:
Locations (1):
- Jones Institute for Reproductive Medicine, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hunzicker-Dunn ME, Lopez-Biladeau B, Law NC, Fiedler SE, Carr DW, Maizels ET. PKA and GAB2 play central roles in the FSH signaling pathway to PI3K and AKT in ovarian granulosa cells. Proc Natl Acad Sci U S A. 2012 Oct 30;109(44):E2979-88. doi: 10.1073/pnas.1205661109. Epub 2012 Oct 8. PMID 23045700
- [Background] Santoro N, Randolph JF Jr. Reproductive hormones and the menopause transition. Obstet Gynecol Clin North Am. 2011 Sep;38(3):455-66. doi: 10.1016/j.ogc.2011.05.004. PMID 21961713
- [Background] Bousfield GR, Butnev VY, Butnev VY, Hiromasa Y, Harvey DJ, May JV. Hypo-glycosylated human follicle-stimulating hormone (hFSH(21/18)) is much more active in vitro than fully-glycosylated hFSH (hFSH(24)). Mol Cell Endocrinol. 2014 Feb 15;382(2):989-97. doi: 10.1016/j.mce.2013.11.008. Epub 2013 Dec 1. PMID 24291635
- [Background] Bousfield GR, Butnev VY, Rueda-Santos MA, Brown A, Hall AS, Harvey DJ. Macro- and Micro-heterogeneity in Pituitary and Urinary Follicle-Stimulating Hormone Glycosylation. J Glycomics Lipidomics. 2014;4:1000125. doi: 10.4172/2153-0637.1000125. PMID 25722940
- [Background] Wang H, May J, Butnev V, Shuai B, May JV, Bousfield GR, Kumar TR. Evaluation of in vivo bioactivities of recombinant hypo- (FSH21/18) and fully- (FSH24) glycosylated human FSH glycoforms in Fshb null mice. Mol Cell Endocrinol. 2016 Dec 5;437:224-236. doi: 10.1016/j.mce.2016.08.031. Epub 2016 Aug 22. PMID 27561202
- [Background] Klein NA, Illingworth PJ, Groome NP, McNeilly AS, Battaglia DE, Soules MR. Decreased inhibin B secretion is associated with the monotropic FSH rise in older, ovulatory women: a study of serum and follicular fluid levels of dimeric inhibin A and B in spontaneous menstrual cycles. J Clin Endocrinol Metab. 1996 Jul;81(7):2742-5. doi: 10.1210/jcem.81.7.8675606.
- [Background] Andreasson B, Bostofte E. Influence of 2 mg estradiol-17 beta on circulating FSH, LH, total and unconjugated estradiol levels in post-menopausal women. Acta Obstet Gynecol Scand. 1981;60(6):555-8. doi: 10.3109/00016348109155485. PMID 6801915
- [Background] Bunyavejchevin S, Panthong C, Limpaphayom KK. Serum estradiol and follicle-stimulating hormone levels in Thai women post total abdominal hysterectomy and bilateral oophorectomy using oral 17 beta-estradiol. J Med Assoc Thai. 2002 Jan;85(1):58-62. PMID 12075721
- [Background] Fahraeus L, Larsson-Cohn U. Oestrogens, gonadotrophins and SHBG during oral and cutaneous administration of oestradiol-17 beta to menopausal women. Acta Endocrinol (Copenh). 1982 Dec;101(4):592-6. doi: 10.1530/acta.0.1010592. PMID 6818806
- [Background] Robyn C, Vekemans M. Influence of low dose oestrogen on circulating prolactin. LH and FSH levels in post-menopausal women. Acta Endocrinol (Copenh). 1976 Sep;83(1):9-14. doi: 10.1530/acta.0.0830009. PMID 989226
- [Background] Wide L, Naessen T. 17 beta-oestradiol counteracts the formation of the more acidic isoforms of follicle-stimulating hormone and luteinizing hormone after menopause. Clin Endocrinol (Oxf). 1994 Jun;40(6):783-9. doi: 10.1111/j.1365-2265.1994.tb02513.x. PMID 8033370
- [Background] Bousfield GR, Butnev VY, Walton WJ, Nguyen VT, Huneidi J, Singh V, Kolli VS, Harvey DJ, Rance NE. All-or-none N-glycosylation in primate follicle-stimulating hormone beta-subunits. Mol Cell Endocrinol. 2007 Jan 2;260-262:40-8. doi: 10.1016/j.mce.2006.02.017. Epub 2006 Oct 31. PMID 17079072
- [Background] Archer DF, Pickar JH, MacAllister DC, Warren MP. Transdermal estradiol gel for the treatment of symptomatic postmenopausal women. Menopause. 2012 Jun;19(6):622-9. doi: 10.1097/gme.0b013e31823b8867. PMID 22282101